CLINICAL TRIAL: NCT03980392
Title: A Randomized Controlled Study to Evaluate Applicability of Korean Multidomain Intervention Program in the South Korean Study to Prevent Cognitive Impairment and Protect Brain Health Through Lifestyle Intervention
Brief Title: South Korean Study to Prevent Cognitive Impairment and Protect Brain Health Through Lifestyle Intervention
Acronym: SUPERBRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor-Investigator, Inha University Hospital, Professor Seong Hye Choi, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HI18C0479
Record Dates: First submitted 2019-05-28; First posted 2019-06-10 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Mild Cognitive Impairment; Aged
Keywords: prevention; dementia; intervention; mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: They will be randomly allocated to facility-based multidomain intervention group, home-based intervention group, and a regular health advice group (referred to as control group) at a ratio of 1:1:1.
Who Masked: Outcomes Assessor
Masking Description: Independent raters are blinded to the group of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facility-based Intervention (Experimental): A group will consist of 5 or 10 persons depending on the size of the study center. Exercise training will be guided by study exercise therapists at a gym and consist of programs for progressive muscle strength training, aerobic exercise, and exercises to improve postural balance and flexibility using elastic bands, floor plate and chairs (three times per week, 60 min per session).The cognitive training program is a program including tasks to be effective in episodic memory, executive function, attention, working memory, calculation, and visuospatial function (twice per week, 60 min per session). The nutritional intervention is conducted by study nutritionists (three individual sessions and seven group sessions). Management of metabolic and vascular risk factors will include additional meetings with the study nurse (at 0, 4, 8, 16, and 20 weeks), and the study physician (at 0 and 12 weeks). Motivational training is conducted by psychologist (four group session).
  Interventions: Other: Multidomain intervention program
- Home-based Intervention (Experimental): The nutritional intervention, management of metabolic and vascular risk factors, social activity, and motivational training in the home-based intervention are similar to the facility-based intervention. The physical exercise programs consist of one group session (60 min) and two home-based sessions (60 min per session) per week in the first 2 months of the trial. During the remaining months of the 6-month study, participants in the home-based intervention attend a 1-h physical exercise group session per two weeks and two or three exercise sessions (60 min per session) alone at home per week. The cognitive training programs consist of one group session (60 min) and one home-based sessions (60 min per session) per week in the first 2 months of the trial. For the remainder of the 6-month study, participants in the home-based intervention attend a 1-h group cognitive training session per two weeks and one or two cognitive training sessions (60 min per session) alone at home per week.
  Interventions: Other: Multidomain intervention program
- Controls (No Intervention): They are waiting list controls. They will receive the multi-domain intervention after this study.

INTERVENTIONS:
Other: Multidomain intervention program — Multidomain intervention program for physical exercise, cognitive training, nutrition, vascular and metabolic risk controls, and motivation
  Arms: Facility-based Intervention; Home-based Intervention

SUMMARY:
This study evaluates acceptability and efficacy of multidomain intervention program to prevent cognitive impairment and protect brain health in Korean at-risk elderly. A third of participants will receive facility-based intervention for 6 months, a third will receive home-based intervention for 6 months, and a third is waiting list controls.

DETAILED DESCRIPTION:
Despite extensive research in the field of Alzheimer's disease (AD), no treatment has yet been developed to modify the progression of AD. Therefore, it is important to manage vascular and metabolic risk factors, to eat healthy foods, to exercise, and to participate in social activities to prevent dementia. The FINGER study showed that the multi-domain intervention program is effective to prevent cognitive impairment and disability in elderly.

In South Korea, exercise and leisure programs, and brain activity for the elderly also have been conducted in welfare centers and public health centers. However, there are not enough programs that have proven effective in the studies.

So the investigators would like to develop a multi-domain intervention program and investigate applicability and efficacy before a large-scale randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 60-79
2. Having at least one among the following dementia risks,

   * hypertension
   * Diabetes Mellitus
   * Dyslipidemia
   * Obesity
   * Abdominal obesity
   * Metabolic syndrome
   * Smoking
   * educational level ≤ 9 years
   * Physical inactivity
   * Social inactivity
3. Independent activities of daily living
4. Mini-Mental State Examination score better than1.5 standard deviations below age and education-adjusted normative means
5. Can read and write Korean
6. Having a reliable informant who could provide investigators with the requested information.
7. Provide written informed consent

Exclusion Criteria:

1. Major psychiatric illness such as major depressive disorders
2. Dementia
3. Substantial cognitive decline
4. Other degenerative disease (e.g., Parkinson's disease)
5. Malignancy within 5 years
6. Cardiac stent or revascularization within 1 year
7. Serious or unstable symptomatic cardiovascular disease
8. Other serious or unstable medical disease such as acute or severe asthma, active gastric ulcer, severe liver disease, or severe renal disease
9. Severe loss of vision, hearing, or communicative disability
10. Any conditions preventing cooperation as judged by the study physician
11. Significant laboratory abnormality that may result in cognitive impairment
12. Unable to participate in exercise program safely
13. Coincident participation in any other intervention trial

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
retention rate (percent) of the participants | 6 months
  Retention rate in each intervention group
compliance (percent) | 6 months
  Compliance to the protocol in each intervention group
Change of cognition | Change at 6 months from baseline
  Repeatable Battery for the Assessment of Neuropsychological Status (sum, range 40-160) / Higher scores mean better cognition.

SECONDARY OUTCOMES:
Change of global cognition | Change at 6 months from baseline
  Mini-Mental State Examination (sum, range 0-30) / Higher scores mean better cognition.
Change of function | Change at 6 months from baseline
  Clinical Dementia Rating scale-Sum of Boxes (sum, range 0-18) / Higher scores mean worse function.
Change of depression | Change at 6 months from baseline
  Geriatric depression scale-15 items (sum, range 0-15) / Higher scores mean worse emotion.
Change of subjective memory complaints | Change at 6 months from baseline
  Prospective and Retrospective Memory Questionnaire (sum, range 18-80) / Higher scores mean worse memory.
Change of memory complaints | Change at 6 months from baseline
  Cognitive Complaint Interview (CCI) (sum, range 0-10) / Higher scores mean worse memory.
Change of prospective memory | Change at 6 months from baseline
  Prospective Memory test (sum, range 0-12) / Higher scores mean better memory.
Change of Quality of life (QOL) | Change at 6 months from baseline
  QOL-Alzheimer's disease (sum, rage 0-52) / Higher scores mean better QOL.
Change of activities of daily livings (ADL) | Change at 6 months from baseline
  Bayer-ADL (averaged, rage 1-10) / Higher scores mean worse ADL.
Change of nutritional status | Change at 6 months from baseline
  Mini Nutritional Assessment (sum, range 0-14) / Higher scores mean better nutrition.
Change of nutrition | Change at 6 months from baseline
  Nutrition Quotient for Elderly (sum, 0-100) / Higher scores mean better nutrition.
Change of balance | Change at 6 months from baseline
  Short Physical Performance Battery (sum, range 0-12) / Higher scores mean better physical function.
Change of physical activity | Change at 6 months from baseline
  Global Physical Activity Questionnaire (This is not scoring.)
Change of motivation | Change at 6 months from baseline
  Motivation Questionnaire subscore 1) Situational Motivation Type Scale (sum, range 4-28) / Higher scores mean better motivation.
  subscore 2) Self-efficacy (sum, range 4-20) / Higher scores mean better motivation.
Adverse event (number of participants) | Up to 24 weeks
  adverse event in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jee Hyang Jeong, MD, PhD, Principal Investigator — Ewha Womans University Hospital; So Young Moon, MD, PhD, Principal Investigator — Ajou University Hospital, Neurology; Chang Hyung Hong, MD, PhD, Principal Investigator — Ajou University Hospital, Psychiatry; Hae Ri Na, MD, PhD, Principal Investigator — Bobath Memorial Hospital; Kyung Won Park, MD, PhD, Principal Investigator — Dong-A University Hospital; Byung Chae Kim, MD, PhD, Principal Investigator — Chonnam National University Hospital; Yoo Kyoung Park, PhD, Study Director — Kyunghee University
Locations (6):
- South Korea (6):
  - Chonnam National University Hospital, Gwangju
  - Inha Univeristy Hospital, Incheon
  - Dong-A University Hospital, Pusan
  - Bobath Memorial Hospital, Seongnam
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No
We will decide it later.

REFERENCES:
- [Derived] Han MH, Lee EH, Park HH, Choi SH, Koh SH. Relationship between telomere shortening and early subjective depressive symptoms and cognitive complaints in older adults. Aging (Albany NY). 2023 Feb 17;15(4):914-931. doi: 10.18632/aging.204533. Epub 2023 Feb 17. PMID 36805537
- [Derived] Park HK, Choi SH, Kim S, Park U, Kang SW, Jeong JH, Moon SY, Hong CH, Song HS, Chun BO, Lee SM, Choi M, Park KW, Kim BC, Cho SH, Na HR, Park YK. Functional brain changes using electroencephalography after a 24-week multidomain intervention program to prevent dementia. Front Aging Neurosci. 2022 Oct 12;14:892590. doi: 10.3389/fnagi.2022.892590. eCollection 2022. PMID 36313025